CLINICAL TRIAL: NCT05824507
Title: The Incidence of Preoperative and Persistent Chronic Endometritis in Women Surgically Treated for Pelvic Endometriosis
Brief Title: Endometriosis and Chronic Endometritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1072.6120.76.2021
Record Dates: First submitted 2023-03-26; First posted 2023-04-21 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Endometriosis; Pelvic Pain; Infertility
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Infertility

STUDY DESIGN:
Intervention Model Description: Prospective cohort tertiary single-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometriosis + empiric antibiotic therapy (Active Comparator): Women undergoing laparoscopic removal of endometriotic foci due to pain/infertility and endometrial aspiration biopsy for diagnosis of CE followed by empirical antibiotic therapy of CE, if confirmed
  Interventions: Diagnostic Test: Endometrial aspiration biopsies for CE diagnosis
- Endometriosis + no empiric antibiotic therapy (Active Comparator): Women undergoing laparoscopic removal of endometriotic foci due to pain/infertility and endometrial aspiration biopsy for diagnosis of CE without empirical antibiotic therapy of CE, if confirmed
  Interventions: Diagnostic Test: Endometrial aspiration biopsies for CE diagnosis

INTERVENTIONS:
Diagnostic Test: Endometrial aspiration biopsies for CE diagnosis — 1 ml of aspirate will be taken from the uterine cavity for histopathological examination and immunohistochemistry for CE during general anesthesia for scheduled surgery

SUMMARY:
Pelvic endometriosis is a complex estrogen-dependent inflammatory syndrome of unknown etiology, altering the microenvironment of the peritoneal cavity and probably endometrial receptivity, and adversely affecting the physiological processes associated with fertilization. Literature data suggest that the distribution of immune system cells in the eutopic endometrium in the presence of endometriosis differs from the physiological state. The functioning of the immune system seems to be significantly modified not only in the foci of endometriosis, but also in the eutopic endometrium, affecting its physiological functions. Chronic endometritis (CE) is a potential factor impairing endometrial receptivity in the course of endometriosis. However, it is not known whether CE is one of the complications of endometriosis or perhaps an element of its pathogenesis. At the moment, endometrial diagnostics is not obligatory in the treatment of endometriosis in women of reproductive age, but it could potentially bring additional benefits and contribute to the improvement of obstetric results and increase the effectiveness of infertility treatment in women with endometriosis.

DETAILED DESCRIPTION:
The aim of the study is:

i) Evaluation of the incidence and activity of CE (expressed as the number of plasma cells / 1 High Power Field, HPF) in women undergoing surgical treatment for pelvic endometriosis due to pain or infertility; ii) Evaluation of the correlation of CE activity (expressed as the number of plasma cells/ 1 HPF) with endometriosis staging according to the American Society for Reproductive Medicine Classification System iii) Evaluation of the impact of surgical removal of pelvic endometriosis foci on CE activity iv) Comparison of the percentage of women with persistent CE after surgery in the subgroup receiving empiric antibiotics (Amoxicillin + Clavulanic Acid 875 mg + 125 mg, twice daily orally for 7 days) and the subgroup without antibiotics. The study will include women aged 18-45 undergoing laparoscopic surgery for pelvic endometriosis. Additionally, an endometrial aspiration biopsy will be performed. Endometriosis will be confirmed by histopathology. The stage of endometriosis will be determined according to revised American Society for Reproductive Medicine Classification. CE will be confirmed by histopathology and immunohistochemical staining with monoclonal murine antibodies against human plasma cells CD138, and will be defined as the presence of plasma cells in the endometrial stroma, the value will be given as the number of plasma cells/1 High Power Field (HPF) and the cut-off will be calculated using the receiver operating characteristic (ROC) curve. A control endometrial biopsy to confirm the effectiveness of empiric antibiotic therapy will be performed up to 3 cycles after the primary procedure.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 years,
* no history of surgical treatment due to reproductive organ pathology,
* no active infection of the genital tract

Exclusion Criteria:

* abdominal surgeries performed within 6 months preceding hospitalization,
* developmental defects of the reproductive organ
* antibiotic or probiotic treatment in the last 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The incidence and activity of CE in study population of women undergoing surgical treatment for pelvic endometriosis due to pain or infertility | up to 3 months
  The number of plasma cells/1 High Power Field (HPF) in endometrial stroma collected by aspiration biopsy determined by immunohistochemistry

SECONDARY OUTCOMES:
The correlation of CE activity with endometriosis stage in study population of women undergoing surgical treatment for pelvic endometriosis due to pain or infertility | up to 3 months
  The correlation between the number of plasma cells/ 1HPF in endometrial stroma and the stage of endometriosis (I-IV) according to the American Society for Reproductive Medicine classification
Comparison of the frequency of persistent CE in the group subjected to postoperative empirical antibiotic therapy and in the untreated group | up to 6 months
  The number of plasma cells/1 High Power Field (HPF) detected by immunohistochemistryin in endometrial stroma collected by aspiration biopsy 3 months after surgery in the group receiving postoperative empiric antibiotic therapy and in the untreated group

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Ph.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Clinic of Gynecological Endocrinology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gawron I, Derbisz K, Jach R, Trojnarska D, Milian-Ciesielska K, Pietrus M. Pelvic peritoneal endometriosis is linked to the endometrial inflammatory profile: a prospective cohort study. BMC Womens Health. 2025 Mar 3;25(1):94. doi: 10.1186/s12905-025-03632-3. PMID 40033263